CLINICAL TRIAL: NCT05852418
Title: Registry Study of the Provision of Assistive Devices, Medicines, and Other Healthcare Measures in an Inter-cohort Observation of Patients With ALS , SMA and Other Neurological Diseases.
Brief Title: Registry Study of Assistive Devices, Medicines and Healthcare Measures in ALS, SMA and Other Neurological Diseases.
Status: Recruiting | Type: Observational
Sponsor: Ambulanzpartner Soziotechnologie APST GmbH (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: EA1/219/15
Record Dates: First submitted 2023-04-28; First posted 2023-05-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS Registry study; SMA Registry study; ALS medication and care registry study; SMA medication and care registry study; NfL; Neurofilament light chain; ALSFRS-R; ALS-App; ALS; APST Research; Biomarker; Tofersen; Nusinersen; Risdiplam
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry study aims to collect data on the provision of assistive devices, medicines, and other healthcare measures, such as ventilation therapy and nutrition support, in patients with Amyotrophic lateral sclerosis (ALS), Spinal muscular atrophy (SMA) and other neurological disorders. The data collected should describe the clinical practice, meaning real-world evidence and patient-reported outcomes.

DETAILED DESCRIPTION:
This registry study aims to collect data on the provision of assistive devices, medicines, and other healthcare measures, such as ventilation therapy and nutrition support, in patients with ALS, SMA and other neurological disorders. The data collected should describe the clinical practice, meaning real-world evidence and patient-reported outcomes. The collected data include clinical characteristics, medical history, assessment scales, such as ALS functional rating scale-revised (ALSFRS-R), prognosis indicators, such as ALS progression rate, biomarker data, such as serum Neurofilament light chain (sNfL), genetic data, such as the mutation status of SOD1, FUS, c9orf72, TARDBP in ALS, SMN1 in SMA patients, innovative drugs such as Tofersen, Nusinersen, Risdiplam, as well as symptomatic drugs, patient-reported outcome data being captured using questionnaires and established clinical scales on medication expectation and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of a chronic neurological disease -

Exclusion Criteria: Lack of cooperation and unwillingness to store and share medical data collected in the registry study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort includes patients with ALS, SMA and other chronic neurological conditions who received care with assistive devices, remedies, medications, or nursing interventions.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2015-10-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The systematic recording of neurological treatment and its evaluation by patients via specific questionnaires | 10 years
  The systematic recording of neurological treatment and its evaluation by patients via specific questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, Prof. Dr., Study Director — Ambulanzpartner Soziotechnologie APST GmbH
Locations (16):
- Germany (16):
  - Christoph Münch, Berlin
  - Neurologische Klinik und Poliklinik, Universitätsklinikum Bergmannsheil, Bochum
  - Klinik für Neurodegenrative Erkrankungen und Gerontopsychiatrie, ALS-Ambulanz und Huntington Ambulanz, Universitätsklinikum, Bonn
  - Klinik und Poliklinik für Neurologie, Medizinische Fakultät Carl Gustav Carus, Technischen Universität Dresden, Dresden
  - Neurologische Klinik, ALS-Ambulanz, Alfried Krupp Krankenhaus Rüttenscheid, Essen, Essen
  - Klinik für Neurologie, Universitätsmedizin, Georg-August-Universität Göttingen, Göttingen
  - ALS- und Muskelambulanz, Medizinische Hochschule Hannover, Hanover
  - Neurologie und Poliklinik, Universitätsklinikum, Heidelberg
  - Ambulanz für Neuromuskuläre und Motoneuron-Erkrankungen, Universitätsklinikum Jena, Jena
  - Klinik und Poliklinik für Neurologie, Leipzig
  - Klinik für Neuroogie-Präzisionsneurologie, Universitätsklinikum Schleswig-Holstein, Universität zu Lübeck, Lübeck
  - Neurologisches Klinik, Ambulanz für Motoneuronerkrankungen und ALS, Diakonissenkrankenhaus, Mannheim
  - Universitätklinikum, Mannheim
  - Klinik und Poliklinik für Neurologie, Klinikum rechts der Isar der Technischen Universität München, München
  - Klinik für Schlafmedizin und Neuromuskuläre Erkrankungen, Westfälische Willhelms-Universität Münster, Münster
  - Klinik für Innere Medizin, Neurologie, UKM Marienhospital Steinfurt, Steinfurt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT05852418/Prot_SAP_000.pdf